CLINICAL TRIAL: NCT01152879
Title: An Evaluation of Quality of Life Outcomes in Cancer Patients Receiving Home Parenteral
Brief Title: Home Parenteral Nutrition in Cancer Patients
Status: Completed | Type: Observational
Sponsor: Southwestern Regional Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: SRMC 10-03
Record Dates: First submitted 2010-06-24; First posted 2010-06-29 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Cancer
Keywords: Parenteral Nutrition; Quality of Life
MeSH Terms: conditions — Neoplasms; Hyperphagia | interventions — Parenteral Nutrition, Home

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Home Parenteral Nutrition: Patients receiving home parenteral nutrition
  Interventions: Dietary Supplement: Home Parenteral Nutrition

INTERVENTIONS:
Dietary Supplement: Home Parenteral Nutrition — Cancer Patients who are discharged on HPN will be monitored for quality of life, nutrition status, pain and nausea medication usage
  Other Names: Intravenous nutrition

SUMMARY:
This study is being done to examine the effect of Parenteral (intravenous) nutrition support in the home setting on quality of life in cancer patients. In addition, this study is being done to examine the effect of home parenteral nutrition on the use of pain and anti-nausea medication.

DETAILED DESCRIPTION:
This is a prospective descriptive non-randomized clinical study to examine quality of life outcomes and use of pain and anti-emetic therapy for patients receiving HPN support. The EORTC QLQ-C30 will be used to evaluate quality of life. All subjects will be monitored monthly throughout the course of treatment for a minimum of 3 months and a maximum of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cancer diagnosis who have been receiving parenteral nutrition in the hospital or have started on HPN while at Cancer Treatment Centers of America and meet the criteria for home parenteral nutrition.
* Patient expected to have a life expectancy of greater than 90 days post discharge.

Exclusion Criteria:

* Patients less than 18 years of age
* HPN patients who do not receive nutrition assessment and follow-up by the Coram Healthcare nutrition support team
* Refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who are candidates for HPN will be identified by the Nutrition and Metabolic Support Team. Patients will be appropriate for HPN as indicated by a safe home environment, readiness for discharge, and reimbursement for the therapy at home. Candidates for HPN include: Patients will a nonfunctioning gastrointestinal tract. Patients that are moderately or severely malnourished (SGA B or C) with aniticipated deterioration in nutritional status due to aggressive treatment. Patients who have failured enteral feedings for nutrition support. Patients with life expectancy of greater than 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life | Monthly for a minimum of 3 months to a maximum of 12 months
  To examine the effect of parenteral nutrition support in the home care setting on quality of life as measured by the EORTC QLQ-C30

SECONDARY OUTCOMES:
Pain and nausea medication usage | Monthly for a minumum of 3 months to a maximum of 12 months
  To examine the effect of home parenteral nutrition on the use of pain medication and anti-emetic therapy administered intravenously, subcutaneously, or orally.

CONTACTS AND LOCATIONS:
Overall Officials: Ross Taylor, MD, Principal Investigator — Cancer Treatment Centers of America at Southwestern Regional Medical Center
Locations (1):
- Cancer Treatment Centers of America at Southwestern Regional Medical Center, Tulsa, Oklahoma, United States

REFERENCES:
- See also: Click here for more information about this study — http://cancercenter.com